CLINICAL TRIAL: NCT07241871
Title: Open-Label Post Market Clinical Follow up Investigation to Evaluate the Clinical Performance and Safety / Tolerability of Lactal Gel for Treatment of Bacterial Vaginosis
Brief Title: Performance and Safety of Lactal Gel for Treatment of Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rolf Kullgren AB (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RKU/006920; DRKS00038289 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Vaginosis; medical device; lactic acid
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactal Gel (Experimental): Lactal Gel (Class IIa medical device): one tube daily administered as vaginal gel for 7 consecutive days, before bedtime
  Interventions: Device: Lactal Gel (Class IIa medical device)

INTERVENTIONS:
Device: Lactal Gel (Class IIa medical device) — One tube of Lactal Gel is daily administered for 7 consecutive days, before bedtime (not during menstrual bleeding period).

SUMMARY:
The aim of this study is to find out how well the medical device Lactal Gel works and how safe it is. The product will be used to treat bacterial vaginosis in a group of fifty women aged 18 years or older.

All participants will receive the one-week treatment as part of their usual medical care.

Each participant will have two visits: one at the beginning of the study (the initial assessment) and another at day 11 (the final visit).

During these visits, the doctor will:

* Perform a normal medical check-up
* Diagnose bacterial vaginosis using the Amsel criteria (which include checking vaginal pH, appearance of discharge, odor, and microscopic examination)
* Ask about symptoms such as odor, discomfort, and itching
* Evaluate, together with the patient, how well the treatment is working
* Assess the patient's satisfaction and how easy the product is to use
* Check that the treatment is safe and well tolerated The results of this study will help doctors choose the most effective and safest treatment for bacterial vaginosis.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and effectiveness of Lactal Gel, a new medical device that is administered vaginally for the treatment of bacterial vaginosis (BV). One group of patients aged 18 years or older who have been diagnosed with BV according to the Amsel criteria will be treated with the tested device for one week. This treatment will be in accordance with the instructions for use of the tested device and the standard usual care of the involved center. The administration of any preparations that may influence the study outcome within the previous three weeks (e.g., antibiotics, antimycotics, probiotics) is prohibited. To diagnose BV, the presence of at least three of the following is required:

* pH >4.5;
* increased thin vaginal discharge;
* amine odor when KOH (Potassium Hydroxide) solution is added to vaginal secretions (Whiff test);
* presence of clue cells in wet preparations.

Patients will be visited at baseline and at day 11 ± 2 (final visit).

The primary outcomes are:

* percentage of BV-free subjects at the final visit.
* Amsel criteria total score at the final visit.

Secondary outcomes are the following:

* patient evaluation for subjective odor, discomfort, and itching
* investigator and patient global evaluation of performance
* safety evaluation by collection of adverse events and by a global safety evaluation performed by patient and investigator
* assessment of patient satisfaction and usability of the tested device

If the results of this study are positive, the new medical device under development has the potential to become a valuable tool for gynecologists. It will be useful in cases where antibiotic treatment is not the preferred option for treating bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria: Participation was based upon written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

* Age ≥ 18 years old, including women of non- childbearing potential such as women after menopause, i.e 12 months after last menstruation
* Newly diagnosed BV episode, based on Amsel criteria (Amsel et al., 1983), i.e. presence of three of the following criteria: increased homogeneous thin vaginal discharge; pH of the secretion >4.5; amine odor when potassium hydroxide (KOH) 10% solution is added to a drop of vaginal secretions; presence of clue cells in wet preparations.
* Suffering from symptoms associated with BV, such as unusual vaginal discharge, odour and discomfort
* Having access to a smartphone or a computer with an internet access and familiar with the use thereof
* to use the Investigational Medical Device (IMD) as recommended (in particular, for 7 consecutive days during the non-bleeding period of the menstrual cycle)
* to avoid the use of any other interventional options for BV during the study (other than the IMD)
* to avoid the use of any other intravaginal product (e.g. suppositories, gels, foams, lubricants, disinfectants, chemically based contraceptives etc.) during the study
* to fill in the electronic Diary (eDiary)
* Commitment to use contraception methods (with the exception of those defined in the previous inclusion criterion)
* Readiness not to participate in another clinical study during this study
* Negative pregnancy testing (beta human chorionic gonadotropin test in urine) at baseline visit

Exclusion Criteria:

* Known allergy or hypersensitivity to the components of the IMD (self-reported)
* Manifested or suspected Candida infection or any other vaginal mycosis
* Trichomoniasis
* Urogenital (dipstick testing), anal or rectal infection within the 3 weeks prior to (self-reported) / at baseline
* History of recurrent genital herpes (self-reported)
* Lesions/infections in the vaginal area
* Use of preparations that may influence the study outcome within the last 3 weeks prior to Baseline and during the study (e.g. antibiotics, antimycotics, probiotics, corticosteroids etc.)
* History in the past 6 months prior to baseline or presence of a sexually transmitted disease (self-reported)
* History or presence of any other clinically significant known (self-reported) condition/disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject
* Pregnancy, nursing or within first 3 months post-partum
* History of or current abuse of drugs, alcohol or medication
* Participation in another study during the last 30 days prior to baseline
* Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 50 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Percent of Bacterial Vaginosis (BV)-free subjects | day 11 ± 2 (final visit)
  Percentage of BV-free subjects evaluated by Amsel criteria (at least of 3 of 4 criteria) and score
Amsel parameter total sum | day 11 ± 2 (final visit)
  Change in mean of the total sum of Amsel criteria scored as follows:
  * pH >4.5=1; pH ≤4.5=0
  * increase thin vaginal discharge=1; not increased thin vaginal discharge=0
  * Whiff test positive=1; whiff test negative=0
  * presence of clue cells in wet preparations=1; absence of clue cells in wet preparations=0

SECONDARY OUTCOMES:
Subjective vaginal odor | day 11 ± 2
  Change of subjective vaginal odor evaluated by the patient using Visual Analogue Score (VAS): 0-10 score
Subjective discomfort | day 11 ± 2
  Change of subjective discomfort evaluated by the patient using VAS (0-10 score)
Subjective itching | day 11 ± 2
  Change of subjective itching evaluated by the patient using VAS (0-10 score)
Investigator global evaluation | day 11 ± 2
  Investigator global evaluation of performance using the 4-points scale: 3=very good; 2=good; 1= moderate; 0= poor
Patient global evaluation | day 11 ± 2
  Patient global evaluation of performance using the 4-points scale: 3=very good; 2=good; 1= moderate; 0= poor
Incidence of adverse events | day 11 ± 2
  The incidence of adverse events (AEs), serious adverse events (SAEs), adverse device effects (ADEs), and serious adverse device effects (SADEs) for the tested medical device will be collected by Investigators and analyzed comparing them with the incidence in standard population
Investigator Global Safety Evaluation | day 11 ± 2
  Global safety evaluation performed by Investigator using the 4-points scale: 3=very good; 2=good; 1= moderate; 0= poor
Patient Global Safety Evaluation | day 11 ± 2
  Global safety evaluation performed by the patient using the 4-points scale: 3=very good; 2=good; 1= moderate; 0= poor
Incidence of Deficiencies | day 11 ± 2
  It will be analyzed and calculated comparing it with the already known deficiencies of the tested device

OTHER OUTCOMES:
Usability: patient satisfaction of the device | day 11 ± 2
  The degree of patient satisfaction with the tested device will be evaluated using the 4-points scale: 3=very satisfied; 2= satisfied; 1= moderately satisfied; 0= not satisfied
Usability: easy of use of the device | day 11 ± 2
  The easy of use of the tested device will be evaluated by the patient using the 5-points scale: 4=very easy; 3= easy; 2= neutral; 1= difficult; 0= very difficult
Usability: willingness to use the device in the future | day 11 ± 2
  Evaluation performed by the patient using the 3-points scale: 2=yes; 1= possibly; 0= no

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Bünemann-Buschmann, Dr. med, Principal Investigator — Frauenarztpraxis Berlin Gemeinschaftspraxis
Locations (1):
- Frauenarztpraxis Berlin Gemeinschaftspraxis, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: The data that support the findings of this study will be available from the corresponding author, upon reasonable request after the result publication.
Access Criteria: The data supporting the findings of this study will be made available to other researchers upon reasonable request from the corresponding author.